CLINICAL TRIAL: NCT06381986
Title: A Clinical Study on the Safety and Efficacy of SHJ002 Sterile Ophthalmic Solution in the Treatment of Corneal Erosion in Patients With Sjogren's Syndrome
Brief Title: Efficacy and Safety of SHJ002 Ophthalmic Solution in the Treatment of Corneal Erosion in Sjogren's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunhawk Vision Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHJ002-SJP2
Record Dates: First submitted 2024-04-12; First posted 2024-04-24 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Corneal Erosion
Keywords: Corneal Erosion

STUDY DESIGN:
Intervention Model Description: Double-Blinded, Parallel, Vehicle-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded, Parallel, Vehicle-Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHJ002 (Experimental): SHJ002 Ophthalmic Solution: topically administered to each eye twice daily for 12 weeks
  Interventions: Drug: SHJ002
- Vehicle (Placebo Comparator): Vehicle: topically administered to each eye twice daily for 12 weeks
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: SHJ002 — Topical ophthalmic
  Arms: SHJ002
Other: Vehicle — Topical ophthalmic
  Arms: Vehicle

SUMMARY:
The purpose of this study is to measure efficacy and safety with 0.25% SHJ002 sterile ophthalmic solution compared to vehicle in treating corneal erosion in Sjogren's patients.

SHJ002 is an antisense oligonucleotide to neutralize a specific microRNA.

DETAILED DESCRIPTION:
Participants will be randomized to treatment with SHJ002 Ophthalmic Solution or vehicle which will be administered to each eye twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older inclusive, at the time of signing the informed consent.
2. Diagnosis with Sjogren's syndrome and have corneal erosion
3. Female participants must be 1 year postmenopausal, surgically sterilized, or females of childbearing potential with a negative urine pregnancy test

Exclusion Criteria:

1. Ocular surface corneal disease, other than corneal erosion and dry eye disease (DED).
2. Lid margin disorder other than meibomian gland dysfunction (MGD)
3. Presence of any ocular condition
4. Any history of eyelid surgery or intraocular/ocular surgery
5. Cauterization of the punctum or punctal plug
6. Use of lid scrubs containing chemicals or baby shampoo, or eyelid makeup
7. Use of any of the contraindicated drugs medications
8. Any changes in the dosing of any chronically used systemic drug
9. Disease, condition, or disorder that in the judgement of Investigator could confound study assessments or limit compliance to study protocol
10. Known history of alcohol and/or drug abuse within 12 months
11. Known allergy or contraindication to any component of investigational product (IP) formulation or diagnostic agents.
12. Participation in any drug or device clinical investigation within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Kaohsiung Medical Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital-Tu Cheng, New Taipei City
  - MacKay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHJ002 | Vehicle
Started | 58 | 58
Completed | 54 | 51
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHJ002 | Vehicle | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.95 (9.43) | 61.12 (10.96) | 61.03 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 58 | 58 | 116
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Total Corneal Fluorescein Staining
Description: The total corneal fluorescein staining score will be assessed using the NEI grading scale (0-15 points; higher scores indicate more severe staining).
Time Frame: Baseline to Week 12
Population: FAS population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SHJ002 | Vehicle
Number analyzed (Participants) | 58 | 58
units on a scale | -2.55 [-3.43 to -1.68] | -0.37 [-1.23 to 0.49]

2. Secondary Outcome: Change From Baseline to Week 12 in Inferior Corneal Fluorescein Staining (iCFS)
Description: iCFS score will be assessed using NEI regional grading (0-3 for the inferior region); higher scores represent more severe staining.
Time Frame: Baseline to Week 12
Population: FAS population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SHJ002 | Vehicle
Number analyzed (Participants) | 58 | 58
score on a scale | -0.79 [-1.07 to -0.52] | -0.14 [-0.41 to 0.13]

3. Secondary Outcome: Change From Baseline to Week 12 in SANDE Score
Description: Symptom Assessment in Dry Eye (SANDE) questionnaire total score, on a 0-100 scale (higher = worse symptoms).
Time Frame: Baseline to Week 12
Population: FAS population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SHJ002 | Vehicle
Number analyzed (Participants) | 58 | 58
score on a scale | -31.21 [-41.21 to -21.21] | -28.87 [-38.15 to -19.59]

ADVERSE EVENTS:
Time Frame: 84 Days
Description: Treatment-emergent adverse event
Arm/Group | SHJ002 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT06381986/Prot_SAP_000.pdf